CLINICAL TRIAL: NCT04024280
Title: Effects of a Physical Exercise Program in Quality of Life of Breast Cancer Survivors
Acronym: MamaMoveGaia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associacao de Investigacao de Cuidados de Suporte em Oncologia (Other)
Collaborators: Centro Hospitalar de Vila Nova de Gaia/Espinho (Other); Aveiro University (Other); University Institute of Maia (Other)
Responsible Party: Principal Investigator, Ana Joaquim, Principal investigator, Associacao de Investigacao de Cuidados de Suporte em Oncologia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MAMA_MOVE_Gaia After Treatment
Record Dates: First submitted 2019-07-06; First posted 2019-07-18 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer; Quality of Life; Physical Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Patients will perform a supervised physical exercise program specifically developed for breast cancer patients, based on the guidelines of the American College of Sports Medicine. The physical exercise program comprises 3 weekly sessions of 60 minutes each. Each session will involve an initial warm-up with light mobility exercises, followed by resistance and aerobic training and ending with a return to calm phase of light stretching exercises.
  Interventions: Other: Physical exercise program
- Control arm (No Intervention): Patients should maintain the usual physical activity

INTERVENTIONS:
Other: Physical exercise program — Frequency: 3 weekly sessions. Intensity of aerobic training: reporting 12-17 in the Borg scale. Time of aerobic training: 10 minutes in the first and second weeks and then 2 added minutes at each 2 weeks. Type of aerobic training: walking and stepping. Intensity of resistance training: without load in the first week and, then, 15 submaximal repetitions. Time of resistance training: 30 minutes. Type of resistance training: using free weights; the lower body exercises will be squat, leg extension, leg curl and calf raise; the upper body exercises will be frontal and lateral arm raise, chest press, seated row and bicep curl.
  Arms: Intervention arm

SUMMARY:
A 16 weeks 3-weekly supervised and adapted physical exercise program will be applied to breast cancer survivors in surveillance and, in estrogen receptor positive cases, under hormonotherapy. The program will be applied in group classes of 20 participants, in the facilities of one local gymnasium, by fitness instructors included in the investigation team. Investigators will evaluate the Health-Related Quality of Life (HRQoL), physical activity, cardiopulmonary fitness, upper limb strength and lower limb functionality. The investigators also aim to evaluate the safety of the program and oncological outcomes such as symptoms related to disease and its treatment and, also, overall survival and disease free survival.

DETAILED DESCRIPTION:
This protocol describes a two-arm prospective non randomized trial that will test the HRQoL effect of a 16 weeks 3-weekly supervised and adapted physical exercise program that combines muscle strength and aerobic training with progressive intensity. The benefits of physical exercise programs in breast cancer survivors is well known. However, the studied programs usually are not generalizable because of needs of specialized exercise professionals and materials. The investigators aim to evaluate if it is possible to obtain the same benefits in HRQoL, physical activity, cardiopulmonary fitness, upper limb strength and lower limb functionality when the program is applied in group classes by trained fitness instructors with exercise strategies based in limited material. Maximum participants of each group class is 20. Each participant will pass through a 16 weeks control phase, during which should maintain the usual physical activity and, then, through a 16 weeks study phase, during which undergoes the physical exercise program. In each phase, the participants will be serially evaluated. During the 32 weeks, each participant will pass through 5 evaluation moments: at baseline, at 8 weeks, at 16 weeks before beginning the study phase, at 8 weeks of physical exercise and 16 weeks of physical exercise at the end of the program. After, investigators aim to evaluate each participant at 3, 6 and 12 months ant, then, yearly.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of breast carcinoma
* Stages 0 to IIIC
* Having undergo primary treatment with curative intent, defined as surgery that can have been complemented with neoadjuvant, or adjuvant, chemotherapy and/or radiotherapy
* Conclusion of the last of the following treatments at least one month before: surgery, chemotherapy or radiotherapy
* At least one consultation in the Medical Oncology Department of the Centro Hospitalar de Vila Nova de Gaia/Espinho
* Assistant medical oncologist consent for the physical exercise practice
* Not meeting the physical activity guidelines of the American College of Sports Medicine (moderate activity ≥ 150 minutes/week ou vigorous activity ≥ 75 minutes/week and ≥ 2 resistance training/week).

Exclusion Criteria:

* Severe anemia (Hb ≤ 8 g/dL)
* Symptomatic moderate anemia (Hb >8 and ≤ 10 g/dL); considered symptoms are: sustained tachycardia, exertion dyspnea, thoracic pain or syncope
* Uncontrolled hypertension
* Uncontrolled diabetes
* Cardiac failure grade >1 in the New York Heart Association evaluation
* History of osteoporosis with Tscore <-2.5 in the lumbar spine and/or femur in the menopause
* Contraindication given by the assistant surgeon

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life | Baseline
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30). This is a patient-reported questionnaire composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100.A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Health Related Quality of Life | Week 8
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30). This is a patient-reported questionnaire composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100.A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Health Related Quality of Life | Week 16
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30). This is a patient-reported questionnaire composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100.A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Health Related Quality of Life | Week 24
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30). This is a patient-reported questionnaire composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100.A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Health Related Quality of Life | Week 32
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30). This is a patient-reported questionnaire composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100.A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Joaquim, MD, Principal Investigator — Centro Hospitalar de Vila Nova de Gaia/Espinho
Locations (1):
- Centro Hospitalar de Vila Nova de Gaia/Espinho, Vila Nova de Gaia, Porto District, Portugal